CLINICAL TRIAL: NCT02832466
Title: Quantifying the Deterioration of Physical Function Along 6 Months in Patients in End Stage Renal Disease
Brief Title: Quantifying the Deterioration of Physical Function in Renal Patients
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Eva Segura Ortí, Professor, Cardenal Herrera University
Other Study IDs: Cardenal Herrera Univeristy
Record Dates: First submitted 2016-07-08; First posted 2016-07-14 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Functional Test — Observation of physical function in hemodialysis patients during a period of 6 months

SUMMARY:
Patients undergoing haemodialysis present a decrease in physical function, but little is known about the rate at which function decreases.

The purpose of this study is quantifying the nature and degree of functional deterioration experienced by stage 5 chronic kidney disease patients during a six month period of maintenance haemodialysis therapy.

ELIGIBILITY:
Inclusion Criteria:

* people under hemodialysis treatment at least 3 months
* be medicable stable
* complete all the physical tests

Exclusion Criteria:

* heart stroke in the previous 6 weeks of the study
* inferior limb amputation without artificial aids
* cerebral vascular disease (ictus, ischemic)
* disability to complete functional tests

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Chronic Kidney Diseases undergoing hemodialysis treatment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Short Physical Performance Battery at 6 months | At the beginning of the study and after 6 months
  Assess lower extremity, which includes objective performance-based measure of balance (side-by-side, semi-tanden and tandem), endurance (4m gait speed) and strength (five chair stands). Each component was scored from 0 to 4 and when summed yielded Short Physical Performance Battery scores between 0 (poor) and 12 (best).
Change from Baseline One Leg Standing Test at 6 months | At the beginning of the study and after 6 months
  Consist in maintain one leg stance for as long as possible. The test was considered normal if the one leg standing time reached 45 seconds.
Change from Baseline Timed Up and Go at 6 months | At the beginning of the study and after 6 months
  To stand up from a standard arms chair, walk 3 meters, turn back the cone walk back and sit down to the chair. The time in seconds is record.
Change from Baseline Sit to Stand to Sit 10 and 60 at 6 months | At the beginning of the study and after 6 months
  For the Sit To Stand 10 participant has to stand up and sit down 10 times and the time needed is record; while for the Sit to stand to sit 60 the participant consist in measures how many repetition the participant can to stand up and sit down during 60 seconds
Change from Baseline On leg heel rise at 6 months | At the beginning of the study and after 6 months
  It measures the strength in the triceps surae in the one leg standing position and has to rise the heel. It measures how many repetitions the participants is can do
Change from Baseline Handgrip strength at 6 months | At the beginning of the study and after 6 months
  To measure the amount of strength developed by each hand in kg
Change from Baseline Six Minutes Walking Time at 6 months | At the beginning of the study and after 6 months
  To walk the longest distance possible in 6 minutes by walking continuously the 20 or 30 metres indicated on the floor. It measures the distance in meters

CONTACTS AND LOCATIONS:
Overall Officials: Eva Segura Ortí, Principal Investigator — Lecturer in the Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Moncada, Valencia, Spain